CLINICAL TRIAL: NCT04093895
Title: A Phase 2 Trial to Evaluate the Safety, Tolerability and Efficacy of PerioSept® (3%) as Adjunct to Scaling and Root Planing in Subjects With Periodontitis
Brief Title: Trial to Evaluate Safety, Tolerability, Efficacy of PerioSept® as Adjunct to SRP in Subjects With Periodontitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Geistlich Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSPD 2
Record Dates: First submitted 2019-09-13; First posted 2019-09-18 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Periodontitis
Keywords: Periodontitis; taurolidine; PerioSept
MeSH Terms: conditions — Periodontitis | interventions — taurolidine

STUDY DESIGN:
Intervention Model Description: single arm, uncontrolled, open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SRP and 3% PerioSept(r) (Experimental): Scaling and root planing followed by 3% PerioSept® drug administration
  Interventions: Drug: PerioSept(r)

INTERVENTIONS:
Drug: PerioSept(r) — Scaling and root planing followed by 3% PerioSept(r) administration
  Other Names: Taurolidine

SUMMARY:
A Phase 2, uncontrolled, open-label, single arm study to evaluate the safety, tolerability and efficacy of PerioSept® (3%) as adjunct to Scaling and Root Planing in subjects with periodontitis.

DETAILED DESCRIPTION:
Open-label, uncontrolled, single arm study to evaluate PerioSept® as adjunct to Scaling and Root Planing in Subjects with moderate to severe Periodontitis.

Up to 12 adult subjects will be enrolled to obtain at least 10 evaluable subjects.

4 study visits will take place for each enrolled subject (V1-V4 within 120 days). An additional optional follow-up visit (V5) at 6 Months might be added later on. On the baseline visit at Day 1 (V2) and if needed Day 2 (V2a) patients will undergo full mouth SRP followed by administration of PerioSept® 3% gel into gingival dental pockets. Treatment of PerioSept® 3% (without SRP) will be repeated at V3.

Eligible subjects must have a minimum of 4 qualifying target teeth defined as a tooth with at least one periodontal pocket with a probing pocket depth (PPD) >= 6mm and bleeding on probing (BOP) at baseline defined as study pockets. All study pockets will be treated with SRP and PerioSept®. Additional teeth identified by investigator as needing SRP per standard of care but not meeting target teeth criteria will be defined as non-target teeth/treatment sites and may also be treated with SRP and PerioSept®.

Dental parameters will only be assessed on the target teeth and each of the 6 sites associated with these teeth (assessment sites). Thus, each eligible patient will have at least 4 Target teeth, a minimum of 4 study pockets and a minimum of 24 assessment sites (6 sites per tooth x 4 target teeth, inclusive of the 4 study pockets) that will be assessed for all study outcome measures.

Overall for all 10 evaluable patients there will be at least 40 target teeth, 40 study pockets and 240 sites for which the study outcome measures will be assessed as specified further below.

Assessments will be conducted over a 12 weeks' and optional 24 weeks' (3 and 6 months respectively) period including safety assessments, assessments of dental parameters (PPD, Clinical attachment level, BOP, recession, Plaque index, Gingival Index) and tolerability assessment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects male or female 18 to 80 years of age, inclusive.
* Subjects must be diagnosed with moderate to severe generalized periodontitis (ADA Classification Case Type III or IV) as determined by the investigator.
* Subjects must have at least 4 qualifying target teeth (having a dental pocket with PPD ≥ 6mm and BOP) (teeth having no endodontic disease - treated or untreated).
* Subjects must have at least 12 teeth in the functional dentition, excluding second and third molars In subjects with limited dentition, tooth loss should not be due to traumatic occlusion
* Females of childbearing potential must agree to use of birth control (hormonal, barrier method or abstinence). Hormonal contraceptives must have started not fewer than 30-days before baseline visit/Day 1.
* Subjects must sign informed consent document(s) prior to initiation of any study-specific procedures and treatments.
* Subjects who are able and willing to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

* History of and/or known risk of life-threatening anaphylactic reactions to taurolidine, any of the components in the investigational drug product.
* Presence of an acute periodontal abscess.
* Subjects with healing disorders (e.g. uncontrolled diabetes mellitus, oral cancer) that could compromise wound healing and/or preclude periodontal surgery.
* Subjects who are taking medications that compromise wound healing presenting with clinical evidence of secondary hyperplastic gingival tissue reactions (e.g. calcium channel blockers or anti-seizure medications)
* Pregnant or nursing female subjects; women of child-bearing potential must have a negative urine pregnancy test.
* Use of systemic antibiotics and, topically applied oral antibiotics and other antimicrobial agents (e.g., chlorhexidine) within 45 days prior to Day 1 or expected use during the study trial period.
* An existing condition that may warrant use of antibiotics during the study trial period.
* Known Human Immunodeficiency Virus infection or other immunodeficiency syndrome.
* Subjects with active infectious diseases (e.g. hepatitis, HIV or tuberculosis)
* Use of agents known to affect periodontal status during the trial and/or use within 45 days prior to Day 1 e.g. immunosuppressants, nasal or oral corticosteroids, calcium channel blockers, phenytoin or anticoagulants.
* Heavy smokers/tobacco users are excluded: defined as those smoking ≥ 10 cigarettes or ≥ 4 cigars or ≥ 4 pipes per day (smokeless nicotine products are NOT excluded)
* Participation in another clinical study with an investigational agent within 90 days prior to Day 1.
* Subjects who received oral health treatments/interventions within 90 days of Day 1, which the investigator believes may interfere with the periodontal parameters to be assessed in this study (e.g., significant dental and/or gum/oral tissue work).
* SRP or periodontal surgery within 12 months prior to Day 1.
* Subject who have a medical and/or dental condition (e.g. a current clinically unstable occlusal situation) and/or use medications/supplements which the investigator believes makes him/her unsuitable for participation in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2020-06-10 (Actual); Study Completion 2020-09-25 (Actual)

PRIMARY OUTCOMES:
Efficacy: Mean probing pocket depth (PPD) reduction (mm) of all study pockets (pockets with PPD > 6 mm and bleeding on probing (BOP) at baseline on target teeth) at subject level and across all subjects | Baseline, Week 12
  Mean probing pocket depth (PPD) reduction (mm) of all study pockets (pockets with PPD > 6 mm and bleeding on probing (BOP) at baseline on target teeth) at subject level and across all subjects

SECONDARY OUTCOMES:
Efficacy: Mean PPD reduction (mm) of all study pockets per patient | Baseline, Week 4
  Mean PPD reduction (mm) of all study pockets per patient
Efficacy: Number of study pockets changing from ≥ 6 mm PPD to ≤5 mm PPD | Baseline; Week 4, 12
  Number of study pockets changing from ≥ 6 mm PPD to ≤5 mm PPD
Efficacy: Change in Clinical attachment level (CAL) of all study pockets | Baseline; Week 4, 12
  Change in CAL of all study pockets
Efficacy: Change in plaque index (PI) of all study pockets | Baseline; Week 4, 12
  Change in PI of all study pockets
Efficacy: Change in gingival index (GI) of all study pockets | Baseline; Week 4, 12
  Change in GI of all study pockets
Efficacy: Change in BOP of all study pockets | Baseline; Week 4, 12
  Change in BOP of all study pockets
Efficacy: Change in recession (REC) of all study pockets | Baseline; Week 4, 12
  Change in REC of all study pockets
Efficacy: Change in PPD of all 6 assessment sites on target teeth | Baseline; Week 4, 12
  Change in PPD of all 6 assessment sites on target teeth
Efficacy: Change in CAL of all 6 assessment sites on target teeth | Baseline; Week 4, 12
  Change in CAL of all 6 assessment sites on target teeth
Efficacy: Change in PI of all 6 assessment sites on target teeth | Baseline; Week 4, 12
  Change in PI of all 6 assessment sites on target teeth
Efficacy: Change in GI of all 6 assessment sites on target teeth | Baseline; Week 4, 12
  Change in GI of all 6 assessment sites on target teeth
Efficacy: Change in BOP of all 6 assessment sites on target teeth | Baseline; Week 4, 12
  Change in BOP of all 6 assessment sites on target teeth
Efficacy: Change in REC of all 6 assessment sites on target teeth | Baseline; Week 4, 12
  Change in REC of all 6 assessment sites on target teeth
Safety/tolerability: Assessment of treatment-emergent adverse events based on dental examination | Day -45 till Month 6
  Assessment of treatment-emergent adverse events based on dental examination
Tolerability: Clinician assessment of local irritation to include assessments of redness/erythema, inflammation/swelling, blisters or erosions, suppuration and other findings at the study treatment pockets or surrounding tissue. | Day 1, 2, 28
  Clinician assessment of local irritation to include assessments of redness/erythema, inflammation/swelling, blisters or erosions, suppuration and other findings at the study treatment pockets or surrounding tissue.
Tolerability: Subject reported tolerability for pain, burning/stinging, sensitivity and taste based on a numeric rating scale | Day 1, 2, 28
  Subject reported tolerability for pain, burning/stinging, sensitivity and taste based on a numeric rating scale

OTHER OUTCOMES:
Exploratory: Clinician reported outcome for delivery device handling and ease of use | Day 1, 2
  Clinician reported outcome for delivery device handling and ease of use
Exploratory: Microbiological counts of periodontal pathogens in biofilm samples of 4 study pockets | Baseline (before treatment); Week 4, 12
  Microbiological counts of periodontal pathogens in biofilm samples of 4 study pockets

CONTACTS AND LOCATIONS:
Overall Officials: Michael McGuire, DDS, Principal Investigator — PerioHealth Clinic Houston
Locations (1):
- Perio Health Professionals, Houston, Texas, United States